CLINICAL TRIAL: NCT05613946
Title: Contrast-enhanced Ultrasound and Shear Wave Elastography for the Treatment of Lymphedema (CASTLE) Study
Brief Title: Contrast-Enhanced Ultrasound and Shear Wave Elastography for the Treatment of Lymphedema
Acronym: CASTLE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christine U. Lee, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-006006
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Lymphedema Arm
Keywords: Lymphaticovenous anastomosis surgery
MeSH Terms: interventions — FS 069; perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Microbubble contrast agent Lumason (Other): While subjects are undergoing standard of operation for arm with lymphedema, the healthy arm will receive intradermal injection of microbubbles and imaged immediately by ultrasound.
  Interventions: Drug: Lumason
- Microbubble contrast agent Optison (Other): While subjects are undergoing standard of operation for arm with lymphedema, the healthy arm will receive intradermal injection of microbubbles and imaged immediately by ultrasound.
  Interventions: Drug: Optison
- Microbubble contrast agent Definity (Other): While subjects are undergoing standard of operation for arm with lymphedema, the healthy arm will receive intradermal injection of microbubbles and imaged immediately by ultrasound.
  Interventions: Drug: Definity

INTERVENTIONS:
Drug: Lumason — Ultrasound microbubble contrast agent intradermal 0.2-0.3 cc of microbubble suspension per injection, 10-12 total injections per upper extremity
  Other Names: sulfur hexafluoride lipid-type A microspheres
  Arms: Microbubble contrast agent Lumason
Drug: Optison — Ultrasound microbubble contrast agent intradermal 0.2-0.3 cc of microbubble suspension per injection, 10-12 total injections per upper extremity
  Other Names: perflutren protein-type A microspheres
  Arms: Microbubble contrast agent Optison
Drug: Definity — Ultrasound microbubble contrast agent intradermal 0.2-0.3 cc of microbubble suspension per injection, 10-12 total injections per upper extremity
  Other Names: perflutren lipid microsphere
  Arms: Microbubble contrast agent Definity

SUMMARY:
The purpose of this research is to determine the preferred microbubble agent (Lumason®, Optison®, and Definity®) for lymphatic channel visualization by ultrasound. This research will also evaluate the utility of preoperative high-frequency B-mode ultrasound with contrast-enhanced ultrasound for presurgical planning, and ultrasound shear wave elastography for assessing treatment response at 6-month follow up.

DETAILED DESCRIPTION:
Part 1 - Evaluate the uptake of microbubble agent (Lumason®, Optison®, and Definity®) for lymphatic visualization by ultrasound.

Part 2 - Combine preoperative high-frequency B-mode ultrasound with contrast-enhanced ultrasound to identify patent lymphatic channels for lymphaticovenous anastomosis presurgical planning. Evaluate the utility of ultrasound shear wave elastography for assessing treatment response at 6-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral lymphedema in the upper extremity (ISL stage 2 or 3) secondary to breast cancer or breast cancer treatment.
* Patient qualifies for LVA surgery as determined by the plastic surgeons performing the surgery (Dr. Bill Tran or Dr. Vahe Fahradyan), and the patient consents to surgery.
* Patient must be able to come to the 6-month clinical follow-up appointment (Part 2 only).
* Patients must be able to understand the study procedures and comply with them for the entire length of the study.
* No contraception is necessary or required.

Exclusion Criteria:

* Pregnant or nursing women.
* Known or suspected hypersensitivity to microbubble contrast agent, perflutren, blood products, albumin, polyethylene glycol (PEG), or egg.31.
* Known or suspected cardiac shunts.
* Prior lymphedema surgery in the upper extremity.
* Tattoo or scar on either upper extremity.
* Current drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent..
* Current or past participation within a specified timeframe in another clinical trial, as warranted by the administration of this intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Lymphatic vessel visualization | 5 minutes after injection
  The time from injection to lymphatic visualization, the duration of contrast visualization, and the longest length of lymphatic channel visualized for each injection site will be determined
High-frequency ultrasound and shear-wave elastography | 1.5 hours for intraoperative CEUS and out-patient SWE both at baseline and 6-month follow-up
  Identify any patent lymphatic channels on CEUS or high-frequency ultrasound that were not detected by the reference standard ICG lymphography. We will additionally measure dermal thickness on B-mode ultrasound and perform SWE at levels comparable to the lymphedema grading metrics routinely collected at surgical visits.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lee, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lymphatic Mapping with Contrast-Enhanced Ultrasound (manuscript) — https://journals.lww.com/prsgo/fulltext/2023/10000/lymphatic_mapping_with_contrast_enhanced.31.aspx